CLINICAL TRIAL: NCT01963780
Title: International Trial to Evaluate the Safety and Effectiveness of The Portable Organ Care System (OCS™) Lung For Recruiting, Preserving and Assessing Expanded Criteria Donor Lungs for Transplantation (EXPAND Trial)
Brief Title: International EXPAND Lung Pivotal Trial
Acronym: EXPANDLung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LUN-012013
Record Dates: First submitted 2013-09-04; First posted 2013-10-16 (Estimated); Results first posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2018-04

CONDITIONS: Lung Transplant
Keywords: lung transplantation; lung preservation; breathing lung transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCS Lung Tx. (Experimental): A prospective, pivotal single arm trial.
  Interventions: Device: OCS Lung Preservation

INTERVENTIONS:
Device: OCS Lung Preservation

SUMMARY:
To evaluate the safety and effectiveness of the OCS™ Lung to recruit, preserve and assess donor lungs that may not meet current standard donor lung acceptance criteria for transplantation.

DETAILED DESCRIPTION:
The OCS™ Lung is to be used to recruit, preserve and assess donor lungs that may not meet current standard donor lung acceptance criteria from one or more of the following characteristics:

* Donor PaO2/FiO2 ≤ 300 mmHg; or
* Expected ischemic time > 6 hours; or
* Donor after Cardiac Death (DCD donor); or
* Donor age ≥55 years old

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following:

  * Donor PaO2/FiO2 ≤ 300 mmHg; or
  * Expected ischemic time > 6 hours; or
  * Donor after Cardiac Death (DCD donor); or
  * Donor age ≥55 years old

Exclusion Criteria:

* • Presence of moderate to severe traumatic lung injury with air and/or blood leak

  * Presence of confirmed active pneumonia or persistent purulent secretions on repeated bronchoscopy evaluation or ET suction
  * Previous history of pulmonary disease
  * Multiple transfusions of >10 pRBCs units
  * ABO incompatibility
  * Tobacco history of >20 pack years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11-22 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Ardehali, MD, Principal Investigator — University of California, Los Angeles; Dirk Van Raemdonck, MD, PhD, Principal Investigator — University of Leuven Medical Center
Locations (11):
- United States (8):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California at Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Emory, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
- University of Leuven Hospital, Leuven, Belgium
- Hannover Medical School, Hanover, Germany
- Hospital Universitario Puerta De Hierro, Madrid, Spain

REFERENCES:
- [Derived] Loor G, Warnecke G, Villavicencio MA, Smith MA, Kukreja J, Ardehali A, Hartwig M, Daneshmand MA, Hertz MI, Huddleston S, Haverich A, Madsen JC, Van Raemdonck D. Portable normothermic ex-vivo lung perfusion, ventilation, and functional assessment with the Organ Care System on donor lung use for transplantation from extended-criteria donors (EXPAND): a single-arm, pivotal trial. Lancet Respir Med. 2019 Nov;7(11):975-984. doi: 10.1016/S2213-2600(19)30200-0. Epub 2019 Aug 1. PMID 31378427

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 93 donor lungs retrieved. 12 excluded for clinical reasons: 6 had contusions or open lung injury resulting in visible air and perfusate leakage into the bronchoalveolar space, 4 had unstable OCS Lung perfusion variables, and persistently low P/F ratio, 1 had persistent oedema, 1 had persistent purulent secretions. 2 were excluded for logistical reasons: 2 patients did not receive a lung transplant because of logistical reasons: 1 was diagnosed with cancer, 1 because no surgeons were available.
Groups:
- Single Arm OCS Lung Transplants: A prospective, pivotal, international single arm trial intended to evaluate the safety and effectiveness of the OCS Lung to recruit, preserve and assess donor lungs that may not meet current standard donor lung acceptance criteria for transplantation.
Period: Overall Study
Arm/Group | Single Arm OCS Lung Transplants
Started | 79 (Patients received lung transplant)
Completed (Subjects completed 12-month follow-up) | 72
Not Completed | 7
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm OCS Lung Transplants
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] — Recipient Age (years)
  years | 55.6 (10.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Donor Age (years)
  years | 47 (16)
Sex: Female, Male [Count of Participants; unit: Participants] — Recipient Sex (Male/Female)
  Participants
    Female | 33
    Male | 46
Sex: Female, Male [Count of Participants; unit: Participants] — Donor Sex (Male/Female)
  Participants
    Female | 33
    Male | 46
Donor Inclusion Criteria [Count of Participants; unit: Participants] — Donor inclusion criteria are defined as age ≥55 years, DCD, expected cross-clamp time >6 hours, or PaO2:FiO2 ≤300 mm Hg.
  Participants
    Age ≥55 years | 22
    DCD | 16
    Expected cross-clamp time >6 h | 11
    PaO2:FiO2 ≤300 mm Hg | 9
    DCD and expected cross-clamp time >6 h | 6
    PaO2:FiO2 ≤300 mm Hg and expected cross-clamp time >6 h | 5
    PaO2:FiO2 ≤300 mm Hg and age ≥55 years | 3
    DCD and age ≥55 years | 3
    DCD and PaO2:FiO2 ≤300 mm Hg | 1
    Expected cross-clamp time >6 h and age ≥55 years | 1
    PaO2:FiO2 ≤300 mm Hg, expected cross-clamp time >6 h, and age ≥55 years | 2
Donor PaO2:FiO2 [Mean (Standard Deviation); unit: mm Hg] — Clinical laboratory value used to assess oxygen status
  mm Hg | 378 (110)
Total cross-clamp time [Mean (Standard Deviation); unit: min] | 609 (127)
Recipient BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.49 (4.6)
Recipient Lung allocation score [Mean (Standard Deviation); unit: score on a scale] — Recipient lung allocation score (LAS) is the value that determines a recipient's urgency on the waitlist. This score is assigned on a scale of 0 to 100, 0 being the least urgent and 100 being the most urgent recipient. Population: Data not available for all recipients
  score on a scale
    number analyzed (Participants) | 70
    (all) | 42.0 (13.5)
Recipient Primary Diagnosis [Count of Participants; unit: Participants]
  Chronic obstructive pulmonary disease or emphysema | 27
  Idiopathic pulmonary fibrosis | 18
  Cystic fibrosis | 12
  Non-specific interstitial pneumonia | 5
  Bronchiectasis | 4
  Sarcoidosis | 2
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Endpoint of Patient Survival at Day-30 Post Transplant and Absence of Primary Graft Dysfunction (PGD) Grade 3 During the First 72 Hours Post Lung Transplant
Description: Primary graft dysfunction is graded on a scale of 0 to 3 according to the 2005 ISHLT PGD grading consensus. Grade 0 is considered the least severe and grade 3 is considered a more severe outcome.
Time Frame: 30 days post lung transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm OCS Lung Transplants
Number analyzed (Participants) | 79
Participants | 43
Statistical Analysis 1: Comparison: Single Arm OCS Lung Transplants; Test type: Superiority — Performance goal is 65%; p = 0.9663, one-sided exact binomial test; Proportion = 0.544, 95% CI 2-sided [0.428 to 0.657]

2. Secondary Outcome: Number of Participants With ISHLT Primary Graft Dysfunction (PGD) Grade 2 or 3 at T72 Hours Post Lung Transplantation
Description: as for outcome 1
Time Frame: 72 hours post lung transplantation
Population: one patient was upgradable at T48 and T72
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm OCS Lung Transplants
Number analyzed (Participants) | 78
Participants | 13
Statistical Analysis 1: Comparison: Single Arm OCS Lung Transplants; Test type: Other — No statistical hypothesis testing; Proportion = 0.167, 95% CI 2-sided [0.092 to 0.268]

3. Secondary Outcome: Number of Participants With Primary Graft Dysfunction Grade 3 at T72 Hours
Description: as for outcome 1
Time Frame: 72 hours post lung transplantation
Population: one patient was ungradable at T48 and T72
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm OCS Lung Transplants
Number analyzed (Participants) | 78
Participants | 5
Statistical Analysis 1: Comparison: Single Arm OCS Lung Transplants; Test type: Other — No statistical hypothesis testing; Proportion = 0.064, 95% CI 2-sided [0.021 to 0.143]

4. Other Pre Specified Outcome: Primary Safety Endpoint: Number of Lung Graft Related Serious Adverse Events During the First 30 Days Post Lung Transplantation
Description: An LGRSAE event is defined as the occurrence of any of the following four categories of adverse events that are also serious; acute rejection, respiratory failure, bronchial anastomotic complication, and major pulmonary-related infection.
Time Frame: 30 days post lung transplantation
Measure: Mean (Standard Deviation); unit: Events per participant
Arm/Group | Single Arm OCS Lung Transplants
Number analyzed (Participants) | 79
Events per participant | 0.3 (0.5)
Statistical Analysis 1: Comparison: Single Arm OCS Lung Transplants; Test type: Other — No statistical hypothesis testing; Mean = 0.3, 95% CI 2-sided [0.1 to 0.4]

5. Other Pre Specified Outcome: Long-term Survival: Survival at 12-months Post-transplant
Description: Survival outcomes were collected through one year post-transplant.
Time Frame: 12-months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm OCS Lung Transplants
Number analyzed (Participants) | 79
Participants | 72

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 30 days post-transplant. Serious adverse events were collected for 30 days post-transplant or through hospital discharge, if longer than 30 days. All-cause mortality was collected for the first 12 months post transplant.
Description: Serious adverse events were collected through regular investigator assessment and/or regular laboratory testing.
Arm/Group | Single Arm OCS Lung Transplants
All-Cause Mortality (participants affected / at risk) | 7/79
Serious Adverse Events (participants affected / at risk) | 61/79
Other Adverse Events (participants affected / at risk) | 67/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm OCS Lung Transplants (N=79)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 28 (31)
Infections and infestations (Infections and infestations) | 27 (38)
Cardiac disorders (Cardiac disorders) | 9 (9)
Renal and urinary disorders (Renal and urinary disorders) | 4 (4)
Vascular disorders (Vascular disorders) | 4 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 16 (18)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Immune system disorders (Immune system disorders) | 2 (2)
Nervous system disorders (Nervous system disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Investigations (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm OCS Lung Transplants (N=79)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders (Cardiac disorders) | 20 (20)
Endocrine disorders (Endocrine disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions (General disorders) | 2 (2)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Immune system disorders (Immune system disorders) | 10 (10)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 19 (21)
Investigations (Investigations) | 4 (4)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Nervous system disorders (Nervous system disorders) | 3 (3)
Psychiatric disorders (Psychiatric disorders) | 6 (6)
Renal and urinary disorders (Renal and urinary disorders) | 8 (8)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 33 (39)
Vascular disorders (Vascular disorders) | 4 (4)
Infections and infestations (Infections and infestations) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall have right to publish results. To balance this right with TransMedics' (TM) proprietary interests, site will submit manuscripts intended for publication for TM's review at least 60d prior to submission date. TM will complete its review within 60d of receipt. TM may request that site delete from its manuscripts any reference to TM confidential information and site shall promptly comply with such request. After 60d period, site will have right to publish manuscript, as amended by TM.